CLINICAL TRIAL: NCT02798302
Title: Preoxygenation With a Bag Valve Mask vs Non-rebreather at Flush Rate
Brief Title: Bag Valve Mask vs Non-rebreather at Flush Rate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hennepin Healthcare Research Institute (Other)
Responsible Party: Principal Investigator, Brian Driver, Associate Research Director, Hennepin Healthcare Research Institute
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Preox-2
Record Dates: First submitted 2016-06-06; First posted 2016-06-14 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Non rebreather (Active Comparator)
  Interventions: Other: Flush rate oxygen using a standard flowmeter (Precision Medical, 8MFA). See description for details. This is specific.
- Bag valve mask without leak (Active Comparator)
  Interventions: Other: Flush rate oxygen using a standard flowmeter (Precision Medical, 8MFA). See description for details. This is specific.
- Bag valve mask with simulated mask leak (Active Comparator)
  Interventions: Other: Flush rate oxygen using a standard flowmeter (Precision Medical, 8MFA). See description for details. This is specific.

INTERVENTIONS:
Other: Flush rate oxygen using a standard flowmeter (Precision Medical, 8MFA). See description for details. This is specific. — A standard oxygen flowmeter will be fully opened and oxygen will be administered for three minutes.

SUMMARY:
Healthy volunteers will participate in a crossover trial comparing preoxygenation with a non-rebreather mask to a bag-valve mask (with and without a simulated mask leak) at the flush rate of oxygen (fully opening standard oxygen flowmeter).

ELIGIBILITY:
Inclusion Criteria:

* Age >17

Exclusion Criteria:

* Pregnant
* Any facial hair more than stubble that might impede a mask seal

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-06; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Fraction of expired oxygen | 3 minutes
  The fraction of expired oxygen will be measured after three minutes of preoxygenation